CLINICAL TRIAL: NCT01116596
Title: Effect of Paracetamol on the Status in Glutathione for the Aged Person
Brief Title: Paracetamol and Glutathion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0072; 2006-006564-36 (EudraCT Number)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Pain; Elderly
Keywords: Glutathione; Paracetamol; elderly people
MeSH Terms: conditions — Chronic Pain | interventions — Acetaminophen

INTERVENTIONS:
Drug: Paracetamol — determine, in subjects aged over 70 years, the blood concentration of glutathione (GSH) and urinary loss of cysteine in the detoxification of paracetamol, when taking paracetamol treatment repeated.

SUMMARY:
Paracetamol is one of the most widely used analgesics in the world especially for chronic pain in the elderly. The metabolism of paracetamol occurs in the liver and involves the use of glutamyl-cysteinyl-glycine (Glutathione (GSH)). Medications such as paracetamol, may reduce the reserves of GSH because it is used for detoxification and elimination. It is well known that the concentration of GSH decrease after administration of paracetamol in humans and animals.

Aging is associated with decreased concentration of GSH in cells and tissues. In the elderly, a decrease of GSH concentration in plasma or red blood cells is associated with decreased physical and mental health.

We wish here to determine, in subjects aged over 70 years, the blood concentration of glutathione (GSH) and urinary loss of cysteine in the detoxification of paracetamol, when taking paracetamol treatment repeated.

DETAILED DESCRIPTION:
Paracetamol is one of the most widely used analgesics in the world especially for chronic pain in the elderly. The metabolism of paracetamol occurs in the liver and involves the use of glutamyl-cysteinyl-glycine (glutathione (GSH)). Medications such as paracetamol, may reduce the reserves of GSH because it is used for detoxification and elimination. It is well known that the concentration of GSH decrease after administration of paracetamol in humans and animals.

Aging is associated with decreased concentration of GSH in cells and tissues. In the elderly, a decrease of GSH concentration in plasma or red blood cells is associated with decreased physical and mental health.

We wish here to determine, in subjects aged over 70 years, the blood concentration of glutathione (GSH) and urinary loss of cysteine in the detoxification of paracetamol, when taking paracetamol treatment repeated.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients over 70 years and treated for over two weeks by oral paracetamol, 3 grams per day (Doliprane ® 1000 mg) as part of their usual care.
* Male and female.

Exclusion Criteria:

* Subject to compliance with the prescribed drug therapy is questionable.
* Subject taking the N-acetyl-cysteine.
* Renal or hepatic disease.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Identify, by determining the concentration of blood GSH how the use of paracetamol at the doses usually prescribed affects the status of GSH

SECONDARY OUTCOMES:
Quantifying the loss of cysteine for detoxification of acetaminophen by measuring the amount of paracetamol cysteine conjugate and mercapturic acid excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France